CLINICAL TRIAL: NCT01065155
Title: Central Blood Pressure and Pulse Wave Velocity: Relationship to Target Organ Damage and Cardiovascular Morbidity-mortality in Diabetic Patients. An Observational Prospective Study. LOD-DIABETES: Study Protocol
Brief Title: Relationship of Central Blood Pressure and Pulse Wave Velocity With Target Organ Damage
Acronym: LOD-DIABETES
Status: Completed | Type: Observational
Sponsor: Fundacion para la Investigacion y Formacion en Ciencias de la Salud (Other)
Responsible Party: Sponsor
Other Study IDs: 428/A/09
Record Dates: First submitted 2010-02-06; First posted 2010-02-09 (Estimated); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Diabetes; Cardiovascular Disease
MeSH Terms: conditions — Diabetes Mellitus; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood and urine).
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Median central blood pressure: Median central blood pressure, lower median group 1 and higher group 2.

SUMMARY:
Diabetic patients show an increased prevalence of non dipping arterial pressure pattern, target organ damage and elevated arterial stiffness. These alterations are associated with increased cardiovascular risk.

The objectives of this study are the following: to evaluate the prognostic value of central arterial pressure and pulse wave velocity in relation to the incidence and outcome of target organ damage and the appearance of cardiovascular episodes (cardiovascular mortality, myocardial infarction, chest pain and stroke) in patients with type 2 diabetes mellitus.

DETAILED DESCRIPTION:
METHODS/DESIGN:

Type of study: This is an observational prospective study with a duration of 5 years, of which the first year corresponds to patient inclusion and initial evaluation, and the remaining four years to follow-up.

Setting: The study will be carried out in the urban primary care setting. Study population: Consecutive sampling will be used to include patients diagnosed with type 2 diabetes between 20-80 years of age. A total of 110 patients meeting all the inclusion criteria and none of the exclusion criteria will be included.

Measurements: Patient age and sex, family and personal history of cardiovascular disease, and cardiovascular risk factors. Height, weight, heart rate and abdominal circumference. Laboratory tests: hemoglobin, lipid profile, creatinine, microalbuminuria, glomerular filtration rate, blood glucose, glycosylated hemoglobin, blood insulin, fibrinogen and high sensitivity C reactive protein. Clinical and 24-hour ambulatory (home) blood pressure monitoring and self-measured blood pressure. Common carotid artery ultrasound for the determination of mean carotid intima-media thickness. Electrocardiogram for assessing left ventricular hypertrophy. Ankle-brachial index. Retinal vascular study based on funduscopy with non-mydriatic retinography and evaluation of pulse wave morphology and pulse wave velocity using the SphygmoCor system. The medication used for diabetes, arterial hypertension and hyperlipidemia will be registered, together with antiplatelet drugs.

DISCUSSION: The results of this study will help to know and quantify the prognostic value of central arterial pressure and pulse wave velocity in relation to the evolution of the subclinical target organ damage markers and the possible incidence of cardiovascular events in patients with type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed of Diabetes Mellitus type 2, and
* aged 20-80 years.

Exclusion Criteria:

* psychological and/or cognitive disorders,
* failure to cooperate,
* educational limitations and problems for understanding written language, failure to sign the informed consent document
* patients participating or who will participate in a clinical trial during the study,
* patients with serious comorbidities representing a threat to life over the subsequent 12 months.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive inclusion will be made of the patients referred to the research unit and who meet the corresponding inclusion criteria, i.e., patients diagnosed with DM2 and aged 20-80 years A total of 52 patients are required in each group, estimating a loss to follow-up of 10%. A final total of 110 patients therefore will be included.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2010-02 (Actual); Primary Completion 2014-02 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Cardiovascular target organ damage (renal, cardiac and vascular) and new cardiovascular events | four years

CONTACTS AND LOCATIONS:
Overall Officials: Manuel A Gomez, MD, Principal Investigator — Fundacion para la investigación y formacion en ciencias de la salud
Locations (1):
- Primary care Research unit. La Alamedilla health centre, Salamanca, Spain

REFERENCES:
- [Derived] Gomez-Marcos MA, Recio-Rodriguez JI, Patino-Alonso MC, Agudo-Conde C, Rodriguez-Sanchez E, Maderuelo-Fernandez JA, Gomez-Sanchez L, Gomez-Sanchez M, Garcia-Ortiz L; LOD-DIABETES Group. Evolution of target organ damage and haemodynamic parameters over 4 years in patients with increased insulin resistance: the LOD-DIABETES prospective observational study. BMJ Open. 2016 Jun 1;6(6):e010400. doi: 10.1136/bmjopen-2015-010400. PMID 27251684
- [Derived] Gomez-Marcos MA, Recio-Rodriguez JI, Gomez-Sanchez L, Agudo-Conde C, Rodriguez-Sanchez E, Maderuelo-Fernandez J, Gomez-Sanchez M, Garcia-Ortiz L; LOD-DIABETES Group. Gender differences in the progression of target organ damage in patients with increased insulin resistance: the LOD-DIABETES study. Cardiovasc Diabetol. 2015 Oct 1;14:132. doi: 10.1186/s12933-015-0293-1. PMID 26427534
- [Derived] Gomez-Marcos MA, Recio-Rodriguez JI, Patino-Alonso MC, Agudo-Conde C, Gomez-Sanchez L, Gomez-Sanchez M, Rodriguez-Sanchez E, Maderuelo-Fernandez JA, Garcia-Ortiz L; LOD-DIABETES Group. Cardio-ankle vascular index is associated with cardiovascular target organ damage and vascular structure and function in patients with diabetes or metabolic syndrome, LOD-DIABETES study: a case series report. Cardiovasc Diabetol. 2015 Jan 16;14:7. doi: 10.1186/s12933-014-0167-y. PMID 25853841
- [Derived] Gomez-Marcos MA, Recio-Rodriguez JI, Rodriguez-Sanchez E, Castano-Sanchez Y, de Cabo-Laso A, Sanchez-Salgado B, Rodriguez-Martin C, Castano-Sanchez C, Gomez-Sanchez L, Garcia-Ortiz L. Central blood pressure and pulse wave velocity: relationship to target organ damage and cardiovascular morbidity-mortality in diabetic patients or metabolic syndrome. An observational prospective study. LOD-DIABETES study protocol. BMC Public Health. 2010 Mar 18;10:143. doi: 10.1186/1471-2458-10-143. PMID 20298558